CLINICAL TRIAL: NCT00668811
Title: Sutent Adjunctive Treatment of Differentiated Thyroid Cancer
Acronym: IIT Sutent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCI-2007-214
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Papillary Thyroid Cancer; Follicular Thyroid Cancer; Differentiated Thyroid Cancer
Keywords: thyroid cancer; metastatic thyroid cancer; differentiated thyroid cancer; papillary thyroid cancer; follicular thyroid cancer; Histologically confirmed; metastatic stage 2,stage 3, or stage 4 differentiated thyroid cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary; Adenocarcinoma, Follicular; Thyroid Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm - Sutent (Experimental): Sutent 37.5 mg/day will be given orally.
  Interventions: Drug: SU011248, Sutent

INTERVENTIONS:
Drug: SU011248, Sutent — Sutent 37.5 mg/day will be given orally after radioactive iodine therapy. Total time of Sutent drug administration will be 52 weeks, absent unacceptable toxicity or disease progression. Sutent is supplied as 12.5mg and 25 mg tablets. Patients are to swallow the tablets whole with approximately 250 ml (8 oz.) of water, fasting each morning. Patients will be given monthly calendars (patient diaries) to document the time when the Sutent pills are taken. At monthly visits, patients will bring back this record and the drug bottles.
  Other Names: Sunitinib

SUMMARY:
This study is comparing a drug called Sutent with standard of care treatment for people with advanced thyroid cancer. Because advanced thyroid cancer is becoming increasingly common and effective treatment options are limited, new therapies are desperately needed.

This study is designed to see if Sutent following therapy with radioactive iodine will target cancer cells and delay disease progression better than standard therapy alone. Newly diagnosed patients, who are scheduled to receive radioactive iodine as part of their standard care are possible candidates. By entering into this study, participants agree to take oral Sutent for approximately two years after completing standard therapy. During this time, study participants will be followed closely by their doctor.

DETAILED DESCRIPTION:
This is a two-stage, phase II, single center, targeted therapy trial enrolling patients with stage 2 (for patients younger than 45 years of age), 3 or 4 differentiated thyroid cancer. The primary objective is to assess progression free survival in this population. Sutent will be given orally at 37.5mg daily for two (2) year, or 26 cycles. Each treatment cycle will consist of 28 days. Upon treatment discontinuation, patients will be followed for survival. The frequency and type of survival follow-up assessments performed will be at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

The study population will consist of men and women with histologically confirmed stage 2 (younger than 45 years of age), 3 or stage 4 differentiated thyroid cancer (e.g., papillary or follicular thyroid cancer) that has been previously treated with at least one course of radioactive iodine therapy and has evidence of residual, recurrent or progressive disease documented by any combination of radiologic studies and thyroglobulin levels.

To be eligible for inclusion, patients must fulfill each of the following criteria:

1. Provide written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
2. Age >18 years.
3. Histologically confirmed stage 2 (younger than 45 years of age), 3 or stage 4 differentiated thyroid cancer (i.e., papillary or follicular thyroid cancer).

   a. If a patient has distant metastases, it must be documented by any combination of radiographic studies or whole body radioiodine scanning.
4. Previously treated with at least one course of radioactive iodine (I-131) therapy.
5. At least one measurable site of disease as defined by the Tumor Assessment Criteria in Appendix 3.
6. Serum thyroglobulin levels inappropriately elevated:

   > 60 ng/mL with thyroid gland > 1 ng/mL without thyroid gland
7. ECOG performance status 0-2.
8. Life expectancy ≥ 3 months.
9. Normal organ function. The definitions of minimum adequacy for organ function required prior to study entry are as follows:

   1. Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) less than or equal to 2.5 x upper limit of normal (ULN), or AST and ALT less than or equal to 5 x ULN if liver function abnormalities are due to underlying malignancy.
   2. Total serum bilirubin less than or equal to 1.5 x ULN.
   3. Serum albumin greater than or equal to 3.0 g/dL.
   4. Absolute neutrophil count (ANC) greater than or equal to 1500/uL.
   5. Platelets greater than or equal to 100,000/uL.
   6. Hemoglobin greater than or equal to 9.0 g/dL
   7. Serum creatinine less than or equal to 1.5 x ULN.
10. Agreement to use contraceptives for women with child bearing potential. Unless surgically sterile, men must agree to use effective contraception during period of therapy.
11. The patient must be aware of the nature of his or her malignancy, understand the protocol requirements, risks, discomforts, and be able and willing to sign an informed consent.

Exclusion Criteria:

Patients who fulfill any of the following criteria will be excluded:

1. Prior systemic chemotherapy or targeted therapy within 3 months prior to enrollment.
2. Prior treatment on a Sutent clinical trial or current treatment on another clinical trial.
3. Prior external beam radiation therapy to the target lesion(s).
4. Life expectancy < 3 months.
5. History of any other carcinomas within the last 5 years, except cured basal cell carcinoma of the skin and cured in-situ cervical cancer.
6. Serious uncontrolled concomitant disease that the Investigator feels might compromise study participation.
7. Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome, or the inability to take oral medication.
8. Any of the following clinical conditions within the 12 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident including transient ischemic attack, pulmonary embolism, ongoing cardiac dysrhythmias of NCI CTCAE grade at least 2, atrial fibrillation of any grade, or QTc interval >450 msec for males or >470 msec for females.
9. Uncontrollable hypertension.
10. Known human immunodeficiency virus infection.
11. Current treatment with therapeutic doses of Coumadin-derivative anticoagulants (low dose Coumadin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
12. Patients with a history of uncontrolled seizures, central nervous system disorders of psychiatric disability judged by the Investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake should be excluded from study.
13. Inability to swallow whole tablets.
14. Unwillingness to participate or inability to comply with the protocol for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-04; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Burman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Britten CD, Kabbinavar F, Hecht JR, Bello CL, Li J, Baum C, Slamon D. A phase I and pharmacokinetic study of sunitinib administered daily for 2 weeks, followed by a 1-week off period. Cancer Chemother Pharmacol. 2008 Mar;61(3):515-24. doi: 10.1007/s00280-007-0498-4. Epub 2007 May 16. PMID 17505827
- [Result] Bikas A, Kundra P, Desale S, Mete M, O'Keefe K, Clark BG, Wray L, Gandhi R, Barett C, Jelinek JS, Wexler JA, Wartofsky L, Burman KD. Phase 2 clinical trial of sunitinib as adjunctive treatment in patients with advanced differentiated thyroid cancer. Eur J Endocrinol. 2016 Mar;174(3):373-80. doi: 10.1530/EJE-15-0930. Epub 2015 Dec 15. PMID 26671977

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm - Sutent
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm - Sutent
Number analyzed (Participants) | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [25 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progressive disease (PD) is defined as unequivocal progression of existing non-target lesions, or the appearance of 1 or more new lesions. Disease progression is accessed using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
Time Frame: 12 months after last patient completes treatment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment Arm - Sutent
Number analyzed (Participants) | 23
days | 241 [114 to 518]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the start of treatment to the time to death from any cause or final data collection, whatever happens first.
Time Frame: 12 months after last patient completes treatment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment Arm - Sutent
Number analyzed (Participants) | 23
days | 1694 [505 to 1898]

ADVERSE EVENTS:
Arm/Group | Treatment Arm - Sutent
All-Cause Mortality (participants affected / at risk) | 23/23
Serious Adverse Events (participants affected / at risk) | 2/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm - Sutent (N=23)
Bowel Obstruction (Gastrointestinal disorders) | 1 (2)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm - Sutent (N=23)
Leukopenia (Blood and lymphatic system disorders) | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Fatigue (General disorders) | 12
Diarrhea (Gastrointestinal disorders) | 12
Muscoskeletal Pain (Musculoskeletal and connective tissue disorders) | 9
Hand-foot Syndrome (Skin and subcutaneous tissue disorders) | 9
Hypertension (Cardiac disorders) | 6
Anemia (Blood and lymphatic system disorders) | 11
Neutropenia (Blood and lymphatic system disorders) | 15
Lymphopenia (Blood and lymphatic system disorders) | 5
Hypopigmentation (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 4
Anorexia (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 7
Heartburn (Gastrointestinal disorders) | 4
Hemorrhoids (Gastrointestinal disorders) | 3
Mucostitis (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 9
Taste Alteration (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 8
GI Hemorrage (Gastrointestinal disorders) | 4
Infection (Infections and infestations) | 4
Increased Alkaline Phosphate (Metabolism and nutrition disorders) | 4
Increased ALT (Metabolism and nutrition disorders) | 11
Increased AST (Metabolism and nutrition disorders) | 11
Increased creatinine (Metabolism and nutrition disorders) | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 6
Proteinuria (Metabolism and nutrition disorders) | 5
GI Pain (Gastrointestinal disorders) | 6
General Pain (General disorders) | 5
Nuerological Pain (Gastrointestinal disorders) | 6
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes